CLINICAL TRIAL: NCT00514462
Title: Instiutional Review Board of Chung Shan Medical University Hospital
Brief Title: Carpal Tunnel Syndrome Treated With 830nm Diode Laser
Acronym: CTS
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chung Shan Medical University (Other)
Collaborators: National Taiwan University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CS07040
Record Dates: First submitted 2007-08-08; First posted 2007-08-10 (Estimated); Last update posted 2007-08-10 (Estimated); Status verified 2007-08

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Lasers, Semiconductor; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): low level laser instrument (Painless Light PL-830, Advanced Chips & Products Crop., USA)
  Interventions: Device: diode laser

INTERVENTIONS:
Device: diode laser — wavelength at 830nm, 9.7J/cm2 for 10 min
  Other Names: Low-level laser

SUMMARY:
The purpose of this study is to determine that 830nm diode laser directly above the transverse carpal ligament (between the pisiform and navicular bone) on subjects' wrists, and test this therapeutic effect.

DETAILED DESCRIPTION:
The low level laser instrument (Painless Light PL-830, Advanced Chips & Products Crop., USA) emitted two light beams with a distance of 2.5cm between them by two laser diodes.

ELIGIBILITY:
Inclusion Criteria:

* no operation of the wrist
* first onset of CTS more than 1 year ago with repeated episodes
* never having laser treatment before.

Exclusion Criteria:

* patients with any rheumatoid arthritis
* history of metabolic disease or paralyzed limbs caused by stroke
* taking any anti-inflammatory drug
* with other treatments, such as acupuncture, physical therapy and wearing orthosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-07; Study Completion 2007-08 (Estimated)

PRIMARY OUTCOMES:
treatment effect | two weeks

SECONDARY OUTCOMES:
EMG, Jamar dynamometer, Carpal tunnel function disability form | two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Ping Han, MD/PhD, Study Director — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University Hospital, Chinese Taipei, Taiwan, China